CLINICAL TRIAL: NCT02130180
Title: Measurement of the Optic Nerve Sheath Diameter by Optic Ultrasound in Diabetic Ketoacidosis and the Relationship to Cerebral Edema
Brief Title: DKA Optic Ultrasound
Acronym: DKA Optic US
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1402-020
Record Dates: First submitted 2014-04-25; First posted 2014-05-05 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-05

CONDITIONS: Diabetic Ketoacidosis; Uncontrolled Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ED T1DM and hyperglycemia without criteria for DKA
- Well controlled T1DM
- ED DKA

SUMMARY:
Diabetic ketoacidosis (DKA) is a complication of type 1, or "insulin-dependent," diabetes (T1DM) and is defined by a high blood glucose level (over 200 mg/dL) coupled with severe acidosis. In this state the body breaks down fat tissue for adequate energy production. This results in ketone and acid production, and ultimately DKA. Cerebral edema (CE), or "brain swelling," can also occur with severe DKA. Current evaluation for DKA-related CE necessitates a high index of clinical suspicion and often times such patients receive advanced brain imaging such as computed tomography (CT) scans.Ocular sonography (ultrasound) is an alternative imaging technique that can provide immediate diagnostic capability at the bedside and minimize radiation exposure. This technique has been used to rapidly and accurately detect increased brain swelling through measurement of the optic nerve sheath diameter (ONSD) in a number of clinical situations including pediatric head trauma, hydrocephalus and ventriculoperitoneal shunt malfunctions, and altitude sickness in adults. Investigators plan to conduct a prospective study including children aged 7-18 years. The objective of this study is to assess the utility of sonographic measurements of the ONSD as a tool for identification of DKA-related CE.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is a complication of type 1, or "insulin-dependent," diabetes (T1DM) and is defined by a high blood glucose level (over 200 mg/dL) coupled with severe acidosis. Children with T1DM lack adequate insulin production. Without insulin, glucose cannot be used by cells to produce energy and blood glucose levels increase. As a result, the body breaks down fat tissue for adequate energy production. This results in ketone and acid production, and ultimately DKA. Often times DKA is present at the time of diabetes diagnosis. Recent estimates suggest that nearly 30% of children that present with DKA are newly diagnosed with diabetes. DKA can also occur as a result of poorly controlled T1DM or poor adherence to insulin therapy. It is common for such patients to have recurrent episodes of DKA, which may lead to permanent brain injury.

Cerebral edema (CE), or "brain swelling," can also occur with severe DKA. It is unclear what causes CE in children with DKA. Proposed mechanisms include changes in blood flow to the brain, inflammatory mediation, and alteration in the intracellular and extracellular fluid composition in the brain. CE can be "clinically apparent" or "subclinical" in terms of symptomatology. Children with clinically apparent DKA-related CE present with neurologic deficits and altered mental status. These children are at risk for herniation of the brain stem due to elevated pressures in and around the brain, and ultimately death. The neurologic manifestations of clinically apparent DKA-related CE typically occur 4-12 hours after the initiation of medical therapy. However, cases have been reported to occur prior to initiation of therapy. Although clinically apparent DKA-related CE is rare, occurring in 0.5-1% of children with DKA, subclinical DKA-related CE is much more common with estimates suggesting that up to 54% of children with DKA have underlying CE that goes clinically undetected. Early identification of both clinically apparent and subclinical DKA-related CE is critical as the time between initial neurologic symptoms and clinical deterioration can be as little as 3 hours. Moreover, early identification of subclinical DKA-related CE may lead to differences in medical therapy.

Current evaluation for DKA-related CE necessitates a high index of clinical suspicion and often times such patients receive advanced brain imaging such as computed tomography (CT) scans. While CT scans can identify CE, this imaging modality exposes patients to ionizing radiation, is expensive, and may take considerable time in some instances. Moreover, CE can occur in the absence of acute change on CT and some patients with subclinical CE may go unidentified. Magnetic resonance imaging (MRI) has been used to identify subclinical DKA-related CE, however this is often time-consuming, expensive, requires sedation, or may be unavailable at some centers. Ocular sonography (ultrasound) is an alternative imaging technique that can provide immediate diagnostic capability at the bedside and minimize radiation exposure. This technique has been used to rapidly and accurately detect increased brain swelling through measurement of the optic nerve sheath diameter (ONSD) in a number of clinical situations including pediatric head trauma, hydrocephalus and ventriculoperitoneal shunt malfunctions, and altitude sickness in adults.

It is believed, no study has used ocular ultrasound to examine the ONSD in the setting of diabetes or DKA for identification of clinically apparent or subclinical CE. It is unclear if patients with T1DM have a fundamentally different baseline ONSD measurement compared to described normal values. It is also unclear how the ONSD varies during times of diabetes-related illness, such as high blood glucose levels without criteria for DKA compared to unequivocal DKA.

Investigators plan to conduct a prospective study including children aged 7-18 years that present to the Children's Endocrinology Clinic and Children's Emergency Department. The objective of this study is to assess the utility of sonographic measurements of the ONSD as a tool for identification of DKA-related CE. Specifically, the primary aim of this study is to measure and compare the mean ONSD in children with well-controlled T1DM to those presenting to the Emergency Department (ED) with DKA and to those presenting to the ED with T1DM and hyperglycemia without criteria for DKA. Investigators hypothesize that the mean ONSD measurement is smaller in children with well-controlled T1DM compared to children presenting to the ED with DKA and compared to children with T1DM and hyperglycemia without criteria for DKA. Secondarily, investigators aim to compare the mean ONSD in children presenting to the ED with DKA to those presenting to the ED with T1DM and hyperglycemia without criteria for DKA. The study team hypothesizes that the mean ONSD measurement is larger in children presenting to the ED with DKA compared children presenting with T1DM and hyperglycemia without criteria for DKA.

ELIGIBILITY:
Inclusion Criteria:

Ages 7-18 years English speaking

DKA group recruited from Children's ED. Criteria for DKA:

1. Hyperglycemia >200 mg/dL AND
2. Venous pH <7.30 AND/OR
3. Bicarbonate level <15 AND
4. Either positive urine or serum ketones

T1DM and hyperglycemia without criteria for DKA (recruited from Children's ED). Criteria for inclusion:

1. Hyperglycemia (>200 mg/dL) not meeting above criteria for DKA

Well-controlled T1DM control group (recruited from Children's Endocrinology Clinic). Criteria for inclusion:

1. Hemoglobin A1c <8% at time of clinic visit
2. No previous episodes of DKA other than at the time of diagnosis
3. Has never had a documented hemoglobin A1c >10%

Exclusion Criteria:

DKA and patients with T1DM and hyperglycemia without criteria for DKA

1. Treatment with more than 10 mL/kg IV fluids prior to transfer from outside hospital
2. Treatment with insulin prior to transfer from outside hospital
3. Patients with type 2 DM
4. Patients with Hyperosmolar Hyperglycemic Nonketotic State
5. Underlying neurologic condition predisposing to changes in ICP (hydrocephalus, ventriculoperitoneal shunt, Chiari I malformation, Chiari II malformation, pseudotumor cerebri, brain tumor)
6. Underlying condition predisposing to changes in intraocular pressure (glaucoma, eye trauma)

Well-controlled T1DM group with poorly controlled disease, defined as:

1. Hemoglobin A1c >8% OR
2. >1 previous episode of DKA, including DKA at time of diagnosis OR
3. Hemoglobin A1c documented >10% any time in the past

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will conduct a cross-sectional study of pediatric patients aged 7-18 years. This study will involve recruitment of patients from both the Endocrinology Clinic and the ED. We will recruit patients from the Children's Endocrinology Clinic with well-controlled T1DM, defined as having a hemoglobin A1c <8% at time of the clinic visit, no previous episodes of DKA other than at the time of diagnosis, and no previous hemoglobin A1c values >10%. This study will also involve recruitment of two subsets of patients from the Children's ED: those with DKA and those with T1DM and hyperglycemia without criteria for DKA.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Mean Optic Nerve Sheath Diameter | 1 day; the day of the ED or clinic visit
  Measure and compare the mean ONSD in children with well-controlled T1DM to those presenting to the ED with DKA and to those presenting to the ED with T1DM and hyperglycemia without criteria for DKA.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bergmann, MS, DO, Principal Investigator — Children's Hospitals and Clinics of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis and Saint Paul, Minnesota, United States